## UNIVERSIDADE FEDERAL DO RIO DE JANEIRO

## AMANDA PEREIRA DA CRUZ



FATORES PREDITIVOS PARA FALHA DA VENTILAÇÃO NÃO-INVASIVA E DA OXIGENOTERAPIA SOB ALTO FLUXO EM PACIENTES COM COVID19: ESTUDO OBSERVACIONAL RETROSPECTIVO

## PESQUISADORES PRINCIPAIS

- Patricia Rieken Macedo Rocco (MD, PhD)
- Cynthia Samary (PhD)
- Fernanda Ferreira Cruz (MD, PhD)
- Amanda Pereira da Cruz (Ft)
- Pedro Leme Silva (PhD)

# **EQUIPE**

## Instituto de Biofísica Carlos Chagas Filho/UFRJ

• Pedro Leme Silva (PhD)

# Instituições Participantes:

- Hospital Barra D'Or
- Laboratório de Investigação Pulmonar, Instituto de Biofísica Carlos Chagas Filho, Universidade Federal do Rio de Janeiro

#### **RESUMO**

Introdução: A COVID-19 é uma doença infecciosa causada pelo SARS-CoV2. Durante a progressão da COVID-19, alguns pacientes podem precisar de ventilação nãoinvasiva (VNI) ou oxigenoterapia por cateter nasal de alto fluxo (CNAF). No entanto, o seu uso tem se mostrado controverso nesta população. Objetivo: Descrever, de forma retrospectiva, possíveis variáveis preditoras relacionadas ao uso da VNI e CNAF, com o intuito de associá-las à sua falha e consequente intubação orotraqueal (IOT). Materiais e Métodos: estudo observacional, retrospectivo, segundo modelo STROBE, a partir da análise de prontuários, entre Março de 2020 e Julho de 2021. Estudo aprovado pelo Comitê Cosubstanciado do IDOR (CAAE: 52534221.5.0000.5249). Critérios de inclusão: maiores de 18 anos, diagnóstico de COVID-19 positivo, internados na UTI do Hospital Barra Dor. Critérios de exclusão: tempo de internação hospitalar menor que 3 dias; pacientes que evoluíram para IOT em tempo menor que 48 horas; pacientes cuja terapia tenha durado menos de 48 horas; pacientes cujo prontuário não tenha as variáveis para o estudo. Desfecho primário: incidência de IOT. Desfechos secundários: tempo para IOT, tempo de internação na UTI e hospitalar e mortalidade intra-hospitalar. Análise estatística: Não houve cálculo amostral devido à natureza exploratória, descritiva e retrospectiva deste estudo. O teste de U de Mann-Whitney será aplicado para avaliar diferenças no tempo de permanência da UTI. O tempo de sobrevivência, assim como tempo de internação hospitalar até o evento serão analisados com estimativas de Kaplan-Meier; o teste de log-rank será utilizado para comparação entre grupos. Os valores de p < 0,05 serão considerados estatisticamente significativos. Resultados preliminares: 82,6% dos prontuários concluíram a fase 1 da coleta de dados. Destes, 64,4% fizeram uso de CNAF, VNI ou ambos. 20% dos prontuários passados pela fase 1 concluíam a fase 2 de coleta, com caracterização da população. A ausência de cardiopatia e demência, assim como o início agudo dos sintomas (menor ou igual à 10 dias) e a idade (entre 40 à 79 anos) demonstraram tendência estatisticamente significativa.

**PALAVRAS-CHAVE**: "COVID-19"; "SARS-CoV-2"; "Síndrome Respiratória Aguda Grave"; "ventilação não-invasiva"; "cateter nasal de alto fluxo"; "Lesão Pulmonar Auto-infligida"; "Unidade de Terapia Intensiva".

#### **ABSTRACT**

Introduction: COVID-19 is an infectious disease caused by SARS-CoV2. During the progression of COVID-19, some patients may require noninvasive ventilation (NIV) or high-flow nasal catheter (CNAF) oxygen therapy. However, its use has proved controversial in this population. Objective: To describe, retrospectively, possible predictor variables related to the use of NIV and CNAF, in order to associate them with their failure and consequent orotracheal intubation (OTI). Materials and Methods: observational, retrospective study, according to strobe model, from the analysis of medical records, between March 2020 and July 2021. Study approved by a cosubstantiated committee of IDOR (CAAE: 52534221.5.0000.5249). Inclusion criteria: over 18 years of age, diagnosis of positive COVID-19, hospitalized in the ICU of Barra Dor Hospital. Exclusion criteria: hospital stay time of less than 3 days; patients who evolved to IOT in less than 48 hours; patients whose therapy (NIV, CNAF or NIV + CNAF) lasted less than 48 hours; patients whose medical records do not have the variables for the study. Primary outcome: incidence of OTI. Secondary outcomes: time for OTI, time of icu and hospital stay and in-hospital mortality. Statistical analysis: There was no sample calculation due to the exploratory, descriptive and retrospective nature of this study. The Mann-Whitney U test will be applied to assess differences in icu length of stay. Survival time as well as hospital stay until the event will be analyzed with Kaplan-Meier estimates; the log-rank test will be used for group comparison. The p-< 0.05 will be considered statistically significant. **Preliminary results**: 82.6% of the medical records completed phase 1 of data collection. Of these, 64.4% used CNAF, NIV or both. 20% of the medical records passed through phase 1 completed phase 2 collection, with characterization of the population. The absence of heart disease and dementia, as well as the acute onset of symptoms (less than or equal to 10 days) and age (between 40 and 79 years) showed a statistically significant trend.

KEY WORDS: "COVID-19"; "SARS-CoV-2"; "Severe Acute Respiratory Syndrome"; "non-invasive ventilation"; "high-flow nasal catheter"; "Self-inflicted Lung Injury"; "Intensive Care Unit."

# LISTA DE FIGURAS E TABELAS

| Figura 1: Linha do tempo, demonstrando as três fases da progressão da COVID-19, | com |
|---|---|
| a associação dos sinais e sintomas | 5 |
| Figura 2: variações da Pes e da Ptp na ventilação passiva, ativa e ativa com prespositiva | |
| Figuras 3: Cardiopatia ou não conforme tratamentos | - 22 |
| Figura 4: Demência ou não, conforme tratamentos | - 22 |
| Figuras 5: Tempo de sintomas, conforme tratamentos | - 23 |
| Figura 6: Faixa etária conforme tratamentos | - 23 |
| Tabela 1:, comorbidades, condição demográfica inicial e tempo de sintomas confo | rme |
| tratamentos utilizadostratamentos utilizados | 21 |
| Tabela 2: Tempo de sintomas e IMC conforme tratamentos utilizados | 21 |

# LISTA DE APÊNDICES

| APÊNDICE 1: Fluxograma de dados preliminares24 |
|------------------------------------------------|
|------------------------------------------------|

## LISTA DE ABREVIAÇÕES E SIGLAS

IRpA – Insuficiência Respiratória Aguda

SARS - síndrome respiratória aguda grave

SAM - síndrome de ativação macrofágica;

SDRA - síndrome do desconforto respiratório agudo

OMS - Organização Mundial da Saúde

ESPII - Emergência de Saúde Pública de Importância Internacional

UTI – unidade de terapia intensiva

SAPS II – Simplified Acute Physiology Score (escore fisiológico agudo simplificado)

DP – dirving pressure (pressão de distensão)

IMC<sup>2</sup> - índice de massa corporal

SRAA – sistema renina-angiotensina-aldosterona

FiO<sub>2</sub> - fração inspirada de oxigênio

PaO<sub>2</sub> - pressão parcial de oxigênio no sangue arterial;

PaO2/FiO2 (P/F) – relação pressão parcial de oxigênio arterial x fração inspirada de oxigênio

PaCO2 – pressão parcial de gás carbônico arterial

pH – potencial hidrogeniônico

HCO3 - bicarbonato

IL - interleucina;

LDH - desidrogenase láctica;

NT-proBNP - porção N-terminal do pró-hormônio do peptídeo natriurético do tipo B;

PCR - proteína C-reativa;

TP - tempo de protrombina.

TGO - transaminase oxalacética

TGP - alanina Aminotransferase

TNF-alfa – fator de necrose tumoral – alfa

IFN-gama – interferon - gama

IP-10 – proteína induzida por interferon gamma 10

ECA-2 – enzima conversora de angiotensina-2

TC – tomografia computadorizada

HD - hemodiálise

SVNI – suporte ventilatório não-invasivo

VMI – ventilação mecânica invasiva

VNI – ventilação não-invasiva

CNAF – cânula nasal de alto fluxo

ECMO – oxigenação por membrana extracorpórea

V/Q – relação ventilação x perfusão

PEEP – pressão positiva expiratória final

P-SILI – patient self-lung injury (lesão pulmonar auto-infligida)

Ppl – pressão pleural

Pes – pressão esofágica

Ptp – pressão transpulmonar

Pva – pressão nas vias aéreas

Vt – *tidal volume* (volume corrente)

CRF – capacidade residual funcional

SpO2 – saturação periférica de O2

FR – frequência respiratória

IPAP – pressão positiva inspiratória

EPAP – pressão positiva expiratória

IOT – intubação orotraqueal

Ang II – angiotensina II

RT-PCR - reação em cadeia da polimerase em tempo real após transcrição reversa

OP – volume de opacidades pulmonares anormais

VPE-TC - volume pulmonar estimado por TC

PPE-TC - peso pulmonar estimado por TC

# ÍNDICE

| 1. | INTRODUÇÃO | 1 |
|---|---|---|
| | 1.1.História e definição da COVID-19 | 1 |
| | 1.2.Epidemiologia da COVID-19 | <b></b> -2 |
| | 1.3.Fisiopatologia da pneumonia por COVID-19 | <b></b> -2 |
| | 1.4.SVNI e oxigenoterapia por CNAF na pneumonia por COVID-19 | <b></b> 7 |
| | 1.5.Possíveis mecanismos de P-SILI na COVID-19 | <b></b> 9 |
| | 1.6.Fatores relacionados à piores desfechos clínicos após SVNI e/ou CNA | ₹F na |
| | pneumonia por COVID-19 | <b></b> 12 |
| 2. | OBJETIVOS | 14 |
| | 2.1. Objetivo geral | 14 |
| | 2.2. Objetivos secundários | 14 |
| 3. | MATERIAIS E MÉTODOS | 15 |
| | 3.1. Delineamento | 15 |
| | 3.2.Local de realização do estudo | 15 |
| | 3.3. Critérios de inclusão | 15 |
| | 3.4. Critérios de exclusão | 15 |
| | 3.5. Fonte de dados | 15 |
| | 3.6. Variáveis coletadas | 16 |
| | 3.7. Análise estatística | <b></b> -17 |
| 4. | ASPECTOS ÉTICOS E DE BOAS PRÁTICAS CLÍNICAS | 18 |
| | 4.1. Aprovação do estudo | <b></b> -18 |
| 5. | DECLARAÇÃO DE CONFIDENCIALIDADE | 18 |
| 6. | ORÇAMENTO | 18 |
| 7. | CRONOGRAMA | 19 |
| 8. | RESULTADOS PRELIMINARES | 20 |
| | 8.1. Análise inicial | 20 |
| 9. | REFERÊNCIAS BIBLIOGRÁFICAS | |

## 1. INTRODUÇÃO

#### 1.1. História e definição da COVID-19

A COVID-19 é uma doença infecciosa, causada pelo vírus SARS-CoV-2, de gravidade variável, acometimento sistêmico (através de agressão viral direta ou por uma resposta inflamatória exacerbada do hospedeiro) e sintomatologia, preferencialmente respiratória, oscilando entre uma síndrome gripal até um quadro respiratório grave, podendo evoluir para a Insuficiência Respiratória Aguda (IRpA) (BERLIN; GULICK; MARTINEZ, 2020a; BOGOCH et al., 2020; HANI et al., 2020; MALIK et al., 2020).

As primeiras notificações surgiram em Wuhan, província de Hubei, na República da China, onde se relatou o surgimento de uma nova cepa de coronavírus, ainda não identificada antes em seres humanos, levando ao crescimento exponencial de uma síndrome gripal atípica, com rápida progressão à um quadro de Síndrome Respiratória Aguda Grave (BOGOCH et al., 2020; https://www.paho.org/pt/brasil - OPAS, acesso em 14 de dezembro de 2021).

Em 30 de Janeiro de 2020, A Organização Mundial de Saúde (OMS) declarou o surto do novo coronavírus uma Emergência de Saúde Pública de Importância Internacional (ESPII), o qual representa o mais alto nível de alerta da Organização, conforme previsto no Regulamento Sanitário Internacional, e dois meses depois, declara a COVID-19 uma pandemia (https://www.who.int/, acesso em 14 de dezembro de 2021).

O primeiro caso de COVID-19 latino-americano foi notificado no Brasil, em Fevereiro de 2020, de um paciente masculino recentemente vindo da Itália, cujo país representou um dos primeiros epicentros da doença no mundo, e um dos primeiros a sofrer um colapso dos seus sistemas de saúde locais (ALBARELLO et al., 2020; <a href="https://www.paho.org/pt/brasil">https://www.paho.org/pt/brasil</a>, acesso em 14 de dezembro de 2021). (RANZANI, et. al. 2021).

A transmissão comunitária no Brasil instalou-se rapidamente, com crescimento exponencial dos casos, internações e mortes, abrindo espaço para as primeiras discussões a respeito das abordagens terapêuticas, principalmente nos casos de IRpA, questionandose a aplicabilidade, eficácia e segurança quanto ao uso de dispositivos

de suporte ventilatório não-invasivo (SVNI) e formas de oxigenoterapia alternativas nos casos de hipoxemia refratária, como o cateter nasal de alto fluxo (CNAF).

#### 1.2. Epidemiologia da COVID-19

Desde seu surgimento, a COVID-19 tem se apresentado como um dos maiores desafios enfrentados pela humanidade em todo período da ciência moderna. Suas características epidemiológicas logo a elencou ao nível pandêmico, levando pesquisadores de todo o mundo a necessidade tangente de desenvolvimento de estudos nas mais diversas áreas, a fim de frear seus impactos de saúde pública e socioeconômicos (OMS, 2021).

A COVID-19 já atingiu aproximadamente 440 milhões pessoas no mundo, levando à 5,9 milhões de pessoas ao morte (https://ourworldindata.org/coronavirus; https://github.com/CSSEGISandData/COVID-19, em Março de 2021 ). No Brasil, até dezembro de 2021, cerca de 29 milhões de pessoas haviam sido diagnosticadas com COVID-19, sendo destas, 650.000 evoluindo para o óbito (https://ourworldindata.org/coronavirus; Ministério da Saúde:https://www.gov.br/pt-br, em Março de 2021).

Um estudo multicêntrico brasileiro observou que, em 2020, 72% dos pacientes internados por COVID-19 necessitaram de algum tipo de suporte ventilatório. Dentre os indivíduos que necessitaram de um leito de terapia intensiva (UTI), aproximadamente 60% morreram e 80% dos ventilados mecanicamente vieram a óbito (RANZANI, *et. al.*,2021).

Em 2021, Kurtz e colaboradores, em um estudo multicêntrico envolvendo 126 UTI's brasileiras, apontaram que, dos pacientes internados na UTI por COVID-19 no período do estudo, 42% evoluíram para IOT e VMI.

A VNI foi utilizada em 37% dos pacientes e, destes, 21% falharam e necessitaram de IOT. O estudo observou que os indivíduos mais jovens, a ausência de condições de fragilidade e o uso de VNI como primeira estratégia de suporte foram independentemente associados ao maior risco de falha (KURTZ, *et. al.*, 2021).

#### 1.3. Fisiopatologia da pneumonia por COVID-19

O SARS-CoV-2 demonstrou, desde o início, grande entropia pelo sistema respiratório, devido às suas características de virulência. Seu mecanismo básico de invasão, através da afinidade de seus receptores *spike* aos receptores das enzimas convertoras de angiotensia 2 (ECA2), presentes em grande quantidade no epitélio respiratório, justificam, em parte, as manifestações clínicas respiratórias observadas (BERLIN; GULICK; MARTINEZ, 2020).

Esta interação dispara a endocitose celular e a fusão da membrana viral com a célula hospedeira, liberando a carga viral no citoplasma do hospedeiro e usurpando o maquinário celular para a produção de novas partículas virais (LOPES-PACHECO et al., 2021; MANCIA et al., 2020).

A replicação e a liberação viral levam a piroptose da célula hospedeira e ativação de vias moleculares associadas ao dano, resultando na liberação de citocinas pró-inflamatórias e quimiocinas. A presença destas citocinas recrutam quimiotaxicamente células do sistema imune adaptativo, com destaque aos linfócitos, que infiltram o tecido pulmonar, podendo explicar, em parte, a linfopenia apresentada em cerca de 80% dos pacientes (TAY et al., 2020).

O desenvolvimento e progressão da COVID-19 apresentam cinco principais mecanismos patológicos, que são: a citotoxicidade viral direta às células que expressam a ECA-2, a desrrregulação do SRAA como resultado da supressão da ECA-2 mediada pelo vírus, a desrregulação do sistema imune, a lesão endotelial e tromboinflamação e a fibrose tecidual como via final do processo inflamatório (LOPES-PACHECO et al., 2021; TAY et al., 2020).

A pneumonia viral é a condição mais observada e o pulmão é o órgão mais vulnerável e afetado pela doença, particularmente pelas vias aéreas possuírem maior expressão dos receptores de ECA-2, além da via de transmissão ser o trato respiratório superior, através da geração e aspiração de aerossóis. O vírus atinge principalmente as células epiteliais das vias aéreas, células epiteliais alveolares, células do endotélio vascular e os macrófagos alveolares (CRUCES et al., 2020; LOPES-PACHECO et al., 2021; RODRIGUEZ-MORALES et al., 2020).

Os achados pulmonares da COVID-19 consistem em dano alveolar difuso e hiperplasia reativa focal dos pneumócitos, com infiltração de células da via inflamatória (principalmente macrófagos e monócitos), vasculite, hipercoagulopatia e trombose

intravascular (BERLIN; GULICK; MARTINEZ, 2020a; RODRIGUEZ-MORALES et al., 2020). Os estudos de análise histopatológica e molecular demonstram grande presença de citocinas pró-inflamatórias no tecido pulmonar, principalmente IL-1, IL-6, TNF-alfa, IFN-gama, IP-10, dentre outras (SIDDIQI; MEHRA, 2020; ZARRILLI et al., 2021).

Como resultado, pode ocorrer colapso alveolar inicial, heterogeneidade pulmonar e mudanças das propriedades viscoelásticas pulmonares, além de alterações micro e macrovasculares, com lesão endotelial vascular e hiperativação da cascata de coagulação por mecanismos tromboembólicos.

Estas alterações levam à um intenso distúrbio da relação ventilação/perfusão (V/Q), com áreas de baixa V/Q e shunt pulmonar (devido à atelectasias, consolidações e preenchimento alveolar por edema exsudativo ricamente proteico) e áreas de alta V/Q e espaço morto fisiológico (devido aos distúrbios da perfusão pulmonar), levando à grandes prejuízos na oxigenação e na mecânica pulmonar (ACKERMANN et al., 2020; BATTAGLINI et al., 2021; ROBBA et al., 2021).

Os sintomas iniciais da COVID-19 são comuns à uma infecção viral, podendo apresentar fadiga, tosse, mialgia, anorexia, febre, dentre outros. Este período podrômico manifesta-se na primeira semana dos sintomas, limitando-se às vias aéreas superiores e evoluíndo, na maioria dos casos, à resolução da doença, (figura 2) (BERLIN; GULICK; MARTINEZ, 2020; LOPES-PACHECO et al., 2021).

No entanto, aproximadamente 15% dos indivíduos acometidos pela COVID-19 irão evoluir para as fases pulmonar e hiperinflamatória, com o desenvolvimento de uma pneumonia de acometimento pulmonar, dispneia e hipoxemia variáveis. Destes, cerca de 5% evoluirão para a forma mais grave, com piora da hipoxemia e rápida progressão para a IrpA (figura 1). (BERLIN; GULICK; MARTINEZ, 2020; LOPES-PACHECO et. al., 2021).



Figura 1: Linha do tempo, demonstrando as três fases da progressão da COVID-19, com a associação dos sinais e sintomas ( Adaptado de Siddiqi HK & Mehra MR. COVID-19 illness in native and imunosupressed states: A clinical-therapeutic staging proposal. J heart Lung Transplant. 2020; 39(5): 405-407).

O diagnóstico pode ser feito a partir da detecção molecular do RNA viral, realizada através de reações de RT-PCR em tempo real (reação em cadeia da polimerase em tempo real após transcrição reversa — síntese de DNA complementar a partir do RNA) (TAHAMTAN; ARDEBILI, 2020). Além disso, a tomografia computadorizada (TC) do tórax também pode proporcionar características que permitem, associada com o quardro clínico e a história natural da doença, diagnosticar e estadiar a COVID-19 (HANI et al., 2020; RODRIGUEZ-MORALES et al., 2020).

Algumas variáveis obtidas pela TC, como a razão entre o volume de opacidades pulmonares anormais e volume pulmonar estimado por TC (VPE-TC) e o peso pulmonar estimado por TC (PPE-TC) podem se correlacionar com a gravidade da pneumonia. Porém, tanto VPE-TC quanto PPE-TC dependem de dados demográficos e variáveis antropométricas (CARVALHO et al., 2021).

Carvalho e colaboradores sugeriram, em 2021, um diagnóstico auxiliado por computador para quantificar a extensão do envolvimento pulmonar em COVID-19, bem como os padrões radiológicos conhecidos como opacidades pulmonares na TC, desenvolvendo um score COVID-19 de gravidade, onde os casos foram classificados como leves (< ponto de corte da normalidade), moderados (ponto de corte da normalidade  $\leq$  3 de envolvimento pulmonar) e envolvimento pulmonar grave (escore  $Z \geq 3$ ) (CARVALHO et al., 2021).

Levando em consideração o alto valor preditivo para a gravidade da COVID-19 que a TC pode proporcionar, estudos futuros podem utilizar os dados de TC de tórax e o grau de comprometimento pulmonar como uma ferramenta capaz de auxiliar na identificação precoce de falha da VNI e/ou CNAF nestes pacientes.

A fim de promover maior entendimento acerca da pneumonia pela COVID-19 e aperfeiçoar as abordagens terapêuticas, foi sugerido a classificação através da progressão do comprometimento pulmonar em três fenótipos: tipo 1 (*Low*), onde se observa opacidades em vidro-fosco multifocais, associado à baixa elastância, baixa V/Q e baixo potencial de recrutabilidade; tipo 2 (intermediário), com aumento das áreas de vidro-fosco, presença de favelamento alveolar, atelectasias e opacidades peribrônquicas, representando a progressão para o tipo 3 (*High*), que é caracterizado pelo estabelecimento de uma forma de SDRA atípica, com intensas áreas de consolidação, atelectasia, preenchimento alveolar, alta elastância e maior potencial de recrutabilidade (GATTINONI et al., 2020; RELLO et al., 2020; ROBBA et al., 2020).

Nas formas mais graves da pneumonia pela COVID-19 a intubação orotraqueal (IOT) e a instituição de ventilação mecainca invasiva (VMI) tornam-se necessárias, com a preconização de ventilação protetora, onde o paciente deve ser ventilado com Vt menor ou igual 6ml/kg de peso predito, pressão de platô igual ou abaixo de 30 cmH<sub>2</sub>O, pressão de distensão (*driving pressure* – DP) igual ou inferior à 15 cmH<sub>2</sub>O, titulação de pressão positiva expiratória final (PEEP) ideal, com hipercapnia e hipoxemia permissivas até limites de segurança (se necessário para manter parâmentros protetores) (BATTAGLINI et al., 2021; BERLIN; GULICK; MARTINEZ, 2020a; MENG et al., 2020).

Com o intuito de melhorar a oxigenação e a mecânica pulmonar nos casos onde o suporte ventilatório invasivo não se encontra suficiente, as terapias de resgate podem ser utilizadas, como o recrutamento alveolar, que consiste na abertura e sua manutenção das unidades alveolares colapsadas, através da aplicação de altos níveis de PEEP de forma decremental, e a posição prona, que através da mudança de decúbito, busca a melhora da distribuição da ventilação das áreas pulmonares posteriores. Se a hipoxemia persistir refratária e o índice de oxigenação (P/F) permanecer igual ou inferior à 150, a oxigenação por membrana extracorpórea (ECMO) é o último recurso (BATTAGLINI et al., 2021; BERLIN; GULICK; MARTINEZ, 2020a; MENG et al., 2020).

#### 1.4. VNI e oxigenoterapia por CNAF na pneumonia por COVID-19

Devido a sua característica de grande transmissibilidade e o crescimento abrupto das formas graves, o impacto significativo nos serviços de saúde e, principalmente, no aumento rápido da taxa de mortalidade, as primeiras recomendações para tratamento da pneumonia por COVID-19 preconizaram a intubação orotraqueal e instalação de VMI como terapia de primeira linha, a fim de evitar a geração de aerossol e evitar a propagação do vírus. Contudo, logo se observou uma alta taxa de mortalidade entre os intubados, além de consumir os recursos e insumos, até então limitados pela crise de saúde pública (BATISTA et al., 2020).

Com o objetivo de proporcionar suporte ventilatório e evitar os impactos negativos advindos da IOT associada à VMI, a VNI e o CNAF adquiriram espaço nos centros de atendimento especializado (FERREYRO et al., 2020; MENG et al., 2020; RISC-19-ICU INVESTIGATORS et al., 2021).

O CNAF é um tipo de oxigenoterapia capaz de ofertar altos níveis de oxigênio sem o ressecamento das vias aéreas superiores, proporcionando maior conforto e melhorando a renovação do gás presente no espaço morto nasofaríngeo.

Atua como um sistema misturador de gás comprimido e oxigênio, administrado através de um cateter nasal de circuito único, fornecendo frações inspiradas de oxigênio (FiO<sub>2</sub>) de até 100% e gerando até 60L/min de fluxo inspiratório de gás aquecido e umedecido, sendo indicada nos casos de IRpA hipoxêmica, a fim de reduzir a necessidade de VNI e VMI (BOCCHILE et al., 2018; NISHIMURA, 2016).

Já a VNI é definida como um suporte de ventilação pulmonar, através de pressão positiva, com o auxílio de interfaces, ou seja, sem o uso de recursos invasivos como intubação traqueal ou traqueostomia, sendo utilizado no suporte inicial da IRpA, nos distúrbios respiratórios agudos, crônicos e crônicos agudizados (XU et al., 2017).

A escolha das interfaces para sua aplicação e sua elegibilidade irão depender do alvo terapêutico, da patologia respiratória (crônica ou aguda) e seu estadiamento, assim como da disponibilidade do dispositivo, do ambiente de aplicação (se domiciliar ou hospitalar) e da experiência do profissional de saúde (ROCHWERG et al., 2017).

Os principais tipos de interface existentes são: 1) os bucais, utilizados por pacientes neuromusculares, em ambiente domiciliar, ofertando um suporte mínimo de pressão positiva, de forma intermitente e sem nenhum tipo de contato contínuo com a pele e

mucosas; 2) as máscaras nasais, que podem ser utilizadas no domicílio ou hospital, proporcionando uma pressão positiva de maior oferta e área de contato mínima da face, além de permite alimentação e fonação. Ela é muito utilizada no tratamento de apnéia obstrutiva do sono, no entanto a perda pressórica pode ser grande se o paciente for um respirador bucal; 3) as máscaras orofaciais, que são as mais utilizadas no ambiente hospitalar nos processos de desconforto respiratório agudo ou crônico-agudizado, ofertando uma pressão positiva de melhor controle, no entanto apresenta maiores pontos de pressão cutânea, não sendo uma opção ideal para períodos prolongados de VNI, além de prejudicar a comunicação e alimentação; 4) as máscaras faciais totais englobam toda a face do indivíduo, proporcionam maior conforto, evitando os pontos de pressão cutânea na ponte do nariz e base dos olhos e permitindo VNI contínua, mas também prejudicam a alimentação e fonação, além de serem mais claustrofóbicas; 5) os capacetes envolvem toda a cabeça do indivíduo, fixando-se com as alças axilares. Evita completamente a face e permite períodos prolongados de VNI, porém também não possibilita alimentação e fonação, além de ser mais complexo e menos acessível na prática clínica (Diretrizes Brasileiras de Ventilacao Mecânica, AMIB-SBPT, Arquivo Eletrônico Oficial, 2013)

De fato, a VNI é um recurso amplamente descrito na literatura, com melhora da oxigenação, redução do desconforto respiratório e melhores desfechos. Entretanto, o seu uso tem se mostrado controverso com relação aos desfechos clínicos nos indivíduos com IRpA e maior acometimento pulmonar por COVID-19. (BERTAINA *et al.*, 2021; RADOVANOVIC *et al.*, 2021; RISC-19-ICU INVESTIGATORS *et al.*, 2021).

Menga e colaboradores (2021) observaram que, entre os pacientes que receberam VNI ou CNAF como terapia de primeira escolha, quando comparados aos pacientes não-COVID-19, apresentaram 2 vezes maior risco de falha. Além disso, dos pacientes COVID-19, 61% que falharam no uso de VNI apresentaram maior risco de mortalidade no curso da internação hospitalar. Os autores sugerem que a alta taxa de mortalidade observada no grupo VNI-COVID-19 pode ser explicada pelo longo período em esforço ventilatório vigoroso, exacerbado pelo aumento da FR e Vt proporcionado pela VNI (MENGA *et al.*, 2021).

Uma revisão sistemática realizada por Radovanovic e colaboradores, em 2021, incluiu 23 estudos retrospectivos, unicêntricos e observacionais prospectivos, que avaliaram falha de VNI/CPAP e mortalidade hospitalar nos pacientes com pneumonia por COVID-19, observaram que, aproximadamente metade destes pacientes evoluíram para

IOT e VMI, e, quando em VMI, a mortalidade chegou a mais de 60% (RADOVANOVIC et al., 2021).

Outros estudos, no entanto, indicam que a VNI em pacientes COVID-19 é um recurso seguro, podendo estar associado à melhores desfechos (BERTAINA et al., 2021; FRANCO et al., 2020; WEERAKKODY et al., 2021). Um estudo multicêntrico transversal do grupo HOPE COVID-19 (2021), que incluiu 36 hospitais em 7 países, realizou uma sub-análise dos pacientes COVID-19 que fizeram uso da VNI, e observou que 37,7% destes pacientes morreram durante a internação e apenas 15% falharam na VNI e/ou CNAF e evoluíram para IOT e VMI (HOPE COVID-19 investigators, 2021).

## 1.5. Possíveis mecanismos da P-SILI na pneumonia por COVID-19

Uma das justificativas para a falha da VNI nesta população é a possível lesão pulmonar auto infligida (P-SILI), gerada pelo esforço muscular respiratório intenso. O aumento do esforço respiratório provoca maior negativação da pressão pleural (Ppl), resultando em maior pressão transpulmonar (Ptp), favorecendo o surgimento de potenciais mecanismos de P-SILI em pacientes com COVID-19 grave (BATTAGLINI *et al.*, 2021; SLUTSKY; RANIERI, 2013).

A P-SILI pode ser definida como a amplificação do dano pulmonar em pulmões previamente lesionados, gerado pela respiração espontânea vigorosa e alto *drive* respiratório, quando a demanda respiratória encontra-se elevada, frente a um processo patológico ou descompensação orgânica (CRUCES et al., 2020; GATTINONI; CARLESSO; CAIRONI, 2012; GRIECO et al., 2019; LIN et al., 2020; SLUTSKY; RANIERI, 2013). Este evento pode ser ainda mais grave quando é aplicada pressão positiva, seja pela VNI ou VMI, sem que haja redução da Ppl e adequação da distribuição da ventilação no intuito de reduzir o esforço respiratório (BATTAGLINI et al., 2021; CRUCES et al., 2020).

Diversos mecanismos fisiopatológicos podem ser sugeridos para a geração de P-SILI nos pacientes COVID-19 sob pressão positiva, onde o aumento do *stress* e o *strain* pulmonar, a heterogeneidade da distribuição da ventilação (*pendelluft*), as alterações da perfusão pulmonar e as assincronias paciente-ventilador mostram-se como os principais mecanismos citados na literatura (BATTAGLINI et al., 2021).

O stress e strain pulmonar se referem aos efeitos biofísicos das pressões e volumes aplicados ao sistema respiratório em cada ciclo respiratório. O stress pulmonar está relacionado a distribuição das forças aplicadas no sistema por unidade de área, ou seja, representa o gradiente pressórico aplicado no sistema respiratório, mais precisamente no componente pulmonar, chamado de pressão transpulmonar (Ptp). Já o strain estima sobredistenção pulmonar e está relacionado ao Vt e ao quanto o pulmão pode se distender a partir da capacidade residual funcional (CRF) (BATTAGLINI et al., 2021; CRUCES et al., 2020; GATTINONI; CARLESSO; CAIRONI, 2012).

Diante de altos esforços inspiratórios, a Ppl torna-se progressivamente mais negativa, gerando altas pressões e volumes pulmonares, que se distribuem heterogenicamente em um pulmão doente. Associado a isto, o perfil de comprometimento pulmonar observado nos pacientes que evoluem para as formas graves de COVID-19 demonstra grandes áreas de heterogeneidade pulmonar, o que resulta em unidades alveolares de diferentes graus de aeração. Isso leva à um prejuízo na oxigenação tecidual, aumentando reflexamente o estímulo respiratório neural. Ambas as situações podem levar à maior negativação da Ppl, com aumento da Ptp e altos Vt, podendo amplificar a P-SILI (BATTAGLINI et al., 2021; GRIECO et al., 2019).

A Pes reflete indiretamente a varaiação da Ppl, e é mensurada através da captação indireta da pressão gerada pela contração diafragmática, transmitida por um cateter esofágico posicionado na porção final do esôfago, próximo ao diafragma. Os pacientes com grande esforço respiratório irão apresentar maior variação da pressão esofágica (Pes). A variação na pressão nas vias aéreas (Pva), seja por respiração espontânea ou por pressão positiva, pode influenciar diretamente na amplitude do *swing* da Pes e, consequentemente, da Ptp. Esta variação é diretamente proporcional aos momentos em que o paciente se encontra em ventilação passiva, ativa e ativa com a pressão positiva. (figura 2) (BATTAGLINI et al., 2021).



Figura 2: variações da Pes e da Ptp na ventilação passiva, ativa e ativa com pressão positiva. (Adaptado de Battaglini et. al. 2021).

A heterogeneidade pulmonar na COVID-19 pode ser explicada pela presença de áreas pulmonares colapsadas, preenchimento alveoar de líquido inflamatório, instabilidade alveolar, com abertura e fechamento cíclico, áreas consolidadas, onde a complacência encontra-se gravemente comprometida e áreas patentes. Essas diferentes áreas desenvolvem, então, diferentes constantes de tempo regionais, resultando em uma distribuição da ventilação alveolar heterogênea, o que pode ser entendido como *pendeluft*, sobredistendento áreas sãs e subexpandindo áreas atelectasicas, principalmente as áreas dependentes pulmonares, resultando em uma insuflação anisotrópica elástica imperfeita (BATTAGLINI et al., 2021; YOSHIDA et al., 2013).

As evidênciais sobre os impactos do *pendeluft* sobre os desfechos e sua aplicabilidade na prática clínica ainda permanecem limitadas, no entanto, considerando o fato de que quanto maior o *pendeluft*, maior o trabalho dispendido para a respiração e que este fenômeno pode ocorrer com considerável frequência (observados em estudos experimentais e observacionais), o *pendeluft* pode ter grande relevância no aumento do risco de desenvolvimento de P-SILI nestes pacientes (BATTAGLINI et al., 2021; GRIECO et al., 2019; YOSHIDA et al., 2013).

Os destúrbios tromboembólicos observados na COVID-19 podem potencializar as alterações da perfusão pulmonar causados pela P-SILI. A tempestade de citocinas

representa um dos principais mecanismos lesivos para o sistema vascular (ROBBA et al., 2020).

O pulmão, já mal perfundido, com grandes áreas de espaço morto fisiológico, ao ser submetido à altos esforços inspiratórios, pode sofrer compressão dos seus capilares, gerando aumento da resistência vascular pulmonar. Além disso, o esforço exacerbado provoca aumento na pressão transcapilar e transalveolar, com lesão de células endoteliais e epiteliais e aumento da perfusão capilar e fluxo sanguíneo locais, podendo resultar em edema e lesão (BATTAGLINI et al., 2021).

A assincronia paciente-ventilador é outro importante mecanismo de P-SILI nos pacientes ventilados mecanicamente. Tanto a subassistência (quando o suporte ventilatório não supre a demanda do paciente), quanto a superassistência (quando o fluxo inspiratório excede a demanda do paciente) podem gerar dissonâncias na ventilação, promovendo maior desconforto ao paciente e alterando a sincronia do tempo neural do paciente e o tempo programado no ventilador. Isto pode favorecer o surgimentos de assincronias secundárias, como as assincronias de ciclagem prematura e duplo-disparos (quando relacionadas à subassistêcia), ou assincronias de ciclagem tardia e disparo ineficaz (nos casos de superassistência) (BATTAGLINI et al., 2021; GRIECO et al., 2019; SLUTSKY; RANIERI, 2013).

Os pacientes com COVID-19 grave apresentam como característica comum o alto drive respiratório. O controle eficaz do esforço respiratório evita lesões diretas e assincronias, prevenindo a P-SILI e a amplificação da lesão pulmonar causada pela VM. Nestes casos a sedação e o bloqueio neuromuscular podem se fazer necessários, a fim de reduzir ou anular, momentaneamente, o estímulo neural exacerbado e assim, promover uma ventilação mais protetora (BATTAGLINI et al., 2021; MENG et al., 2020).

# 1.6. Fatores relacionados à piores desfechos clínicos após Ventilação Não-Invasiva na pneumonia por COVID-19

Os achados relacionados aos desfechos dos pacientes tratados com VNI e/ou CNAF na COVID-19 são incertos e, apesar de haver benefícios observados em alguns estudos, os dados relacionados à morbimortalidade não se mostram muito favoráveis. Weerakkody e

colaboradores, em 2021, observaram em sua revisão de literatura, que reuniu 83 estudos observacionais e 2 ensaios clínicos à respeito dos diferentes dispositivos não invasivos utilizados no suporte ventilatório de pacientes com pneumonia por COVID-19, que, apesar da VNI apresentar-se segura e ser capaz de promover melhores desfechos, esses resultados dependerão de fatores relacionados ao paciente, como a idade avançada, a presença de comorbidades e a gravidade da doença (ALRADDADI et al., 2019; BERTAINA et al., 2021; FRANCO et al., 2020; WEERAKKODY et al., 2021).

Outros fatores de risco multivariáveis para a falha também são citados por Weerakkody, como o grau de hipoxemia no momento da admissão hospitalar, o grau de IrpA antes da instituição da VNI, descrito como SpO<sub>2</sub>/FiO<sub>2</sub>, PaO<sub>2</sub>/FiO<sub>2</sub> ou Índice de ROX ([SpO<sub>2</sub>/FiO<sub>2</sub>]/FR), a pouca melhora na função respiratória após uma tentativa de VNI por 1-6 horas e uma concentração elevada de Proteía C-reativa (PCR).

Já os fatores de risco univariáveis incluíram outros marcadores inflamatórios, o sexo masculino e a FR, mesmo não sendo considerados em alguns estudos como preditores independentes (WEERAKKODY et al., 2021).

A VNI pode, momentâneamente, melhorar a oxigenação e o status clínico sem necessariamente mudar a progressão da doença, dificultando a identificação precoce dos pacientes com alto risco de falha e o momento ideal para IOT. O uso de escalas e preditores de falha validados para a população-alvo podem ser utilizados, com o intuito de auxiliar no seu reconhecimento precoce (BATTAGLINI et al., 2021; MENGA et al., 2021).

Apesar dos dados apresentados, a literatura ainda carece de informações mais robustas a respeito da P-SILI, possivelmente amplificada pela VNI nesta população, enfatizando a necessidade de maior investigação na relação entre: os aspectos relacionados ao uso da VNI e/ou CNAF, como os tipos de interface, os parâmetros ventilatórios ajustados, períodos prolongados na VNI e/ou CNAF, terapias concomitantes (dentre outros fatores) e desfechos clínicos, como dias de internação hospitalar, tempo para falha da VNI e/ou CNAF, com possível indicação de IOT e mortalidade intra-hospitalar.

Este conhecimento pode proporcionar uma identificação mais precoce dos pacientes com potenciais de amplificação da P-SILI frente à VNI e à CNAF e evitar condutas que conduzam à falha desta terapia e suas repercussões.

#### 2. OBJETIVOS

### 2.1. Objetivo geral:

 Descrever, de forma retrospectiva, possíveis variáveis preditoras para a falha da VNI, CNAF ou quando combinadas, e consequente IOT em pacientes com COVID-19 em hospital terciário do Rio de Janeiro.

## 2.2. Objetivos secundários:

- Descrever os tipos de interface de suporte não invasivo [capacete, facial total, oronasal e (cateter nasal de alto fluxo)], assim como os parâmetros ventilatórios utilizados;
- Identificar o uso ou não de oxigênio (sem necessidade, até 1 LO<sub>2</sub>/min, de 1 a 5 LO<sub>2</sub>/min e maior que 5 LO<sub>2</sub>/min) dos pacientes submetidos à VNI, CNAF ou VNI + CNAF, durante e após o uso do dispositivo;
- Identificar se o uso concomitante de alguns medicamentos, como corticosteróides e anticoagulantes, poderiam estar relacionados aos desfechos clínicos;
- Identificar os pacientes que evoluíram para terapia de hemodiálise durante o curso do estudo como uma forma de inferir danos distais;
- Identificar desfechos clínicos relacionados a incidência de IOT (falha da VNI e/ou CNAF), assim como o tempo para IOT, tempo de internação na UTI e hospitalar e mortalidade intra-hospitalar;
- Comparar os pacientes que fizeram uso da VNI sob altos volumes correntes (Vt > 6ml/por Kg peso predito) com aqueles que realizaram a mesma terapia sob baixos volumes correntes (Vt </= 6ml/kg peso predito) ou os níveis de pressão nas vias aéreas (Pva > 15cmH2O ou </= 15cmH2O, respectivamente), assim como no tempo de uso da VNI e/ou CNAF (VNI (3-5 dias, 5-7 dias e > 7 dias), a fim de buscar inferências sobre esforços musculares vigorosos e piores desfechos clínicos;
- Observar se há associação de piores desfechos clínicos em VNI e/ou CNAF de acordo com o grau de acometimento pulmonar através da TC de tórax (menor que 25%; entre 25 e 50% e maior que 50% de área acometida) no momento de admissão hospitalar.

#### 3. MATERIAIS E MÉTODOS

#### 3.1. Delineamento:

Estudo unicêntrico, observacional retrospectivo. O estudo será conduzido de acordo com o *Strengthening the Reporting of Observational Studies in Epidemiology (STROBE):* Explanation and Elaboration (VON ELM, et al., 2007).

### 3.2. Local de realização do estudo:

Será realizado na unidade de terapia intensiva de um hospital terciário, localizado no Rio de Janeiro, RJ.

#### 3.3. Critérios de inclusão:

Pacientes adultos, maiores de 18 anos, internados na UTI com COVID-19 confirmado através de RT-PCR positivo ou TC de tórax sugestiva de pneumonia causada por COVID-19, admitidos entre Março de 2020 e Julho de 2021.

#### 3.4. Critérios de exclusão:

- Tempo estimado de internação hospitalar menor que 3 dias;
- Pacientes que evoluíram para IOT em tempo menor que 48 horas de internação hospitalar;
- Pacientes cujo uso da VNI e/ou CNAF tenha durado menos de 48 horas;
- Pacientes cujo prontuário esteja ausente de variáveis preditivas e de desfecho.

#### 3.5. Fonte de dados:

Os dados serão coletados a partir de prontuários eletrônicos como parte dos cuidados de rotina da UTI. O acesso aos dados será gerenciado pelo centro coordenador da administração hospitalar e disponibilizado aos autores deste projeto, como uma lista, onde constarão todos os pacientes internados no período proposto do estudo e com diagnóstico

positivo para a COVID-19. A partir desta lista, será autorizado o acesso aos respectivos prontuários.

#### 3.6. Variáveis coletadas:

- Admissão hospitalar: tempo do início dos sintomas (em dias), diagnóstico de RT-PCR positivo para COVID-19 ou por TC sugestiva de pneumonia causada por COVID-19, comorbidades (Diabetes melitus, hipertensão arterial sistêmica, doença cerebrovascular, cardiopatias, obesidade, doença pulmonar obstrutiva crônica, asma, pneumopatias estruturais, uso crônico de corticoterapia, doença renal crônica, imunossuprimidos), exames laboratoriais ((D-dímero, PCR, leucócitos, linfócitos, TGO, TGP, bilirrubinna e plaquetas), dados demográficos (idade, gênero, peso, altura, IMC²), uso de medicamentos pré-internação e escores prognósticos (escore SAPS II, probabilidade de óbito [equação geral], Charlson);
- <u>Variáveis preditoras ventilatórias</u>: relacionadas aos dispositivos (tipo de interface, modo e duração em dias) e variáveis ventilatórias (volume corrente, frequência respiratória, saturação periférica de O<sub>2</sub>) e gasométricas (pH, PaO<sub>2</sub>, PaCO<sub>2</sub> e HCO<sub>3</sub> e lactato);

  <u>Nota</u>: As gasometrias serão registradas da seguinte forma: a primeira gasometria coletada a partir da admissão hospitalar e a última na iminência da IOT (em caso de falha da VNI e/ou CNAF) ou a última coletada até o desmame completo e alta hospitalar (em caso de sucesso do VNI e ou CNAF);
- <u>Variáveis preditoras relacionadas as terapias concomitantes</u> (uso de corticosteróides e anticoagulantes) que possam estar relacionados aos desfechos clínicos;
- Variáveis de desfecho clínico:
  - Primário: taxa de intubação orotraqueal e início de ventilação mecânica invasiva;
  - <u>Secundários:</u> 1) necessidade de oxigênio suplementar (sem necessidade, até 1 LO<sub>2</sub>/min, de 1 a 5 LO<sub>2</sub>/min e maior que 5 LO<sub>2</sub>/min, ou porcentagem no caso do CNAF) ao longo da aplicação da terapia; 2) taxa de pacientes que evoluíram para terapia de hemodiálise durante a internação hospitalar; 3) tempo de internação na UTI e hospitalar e taxa de mortalidade intra-hospitalar;
- Os dados coletados e os resultados das inferências propostas nos objetivos secundários deste projeto serão organizados e categorizados em duas tabelas. A primeira tabela estará relacionada aos dados demográficos, como: gênero, idade, peso, altura, IMC<sup>2</sup>,

comorbidades, escore SAPS II (escore prognóstico) e dados coletados no momento da admissão do paciente. A segunda tabela estará relacionada aos dados clínicos e laboratoriais dos pacientes submetidos à VNI e/ou CNAF, sendo:

- Exames laboratoriais (D-dímero da admissão, maior da internação e de alta; PCR de admissão, maior da internação e da alta; leucócitos, linfócitos, TGO e TGP da admissão, a maior da internação e de alta; bilirrubinna de admissão, maior da internação e da alta; plaquetas da admissão, maior dosagem da internação e de alta);
- TC de tórax (com porcentagem de acometimento pulmonar e tipo de vidro fosco);
- Relação PaO<sub>2</sub>/FiO<sub>2</sub>, gasometria arterial (PaO<sub>2</sub>, PaCO<sub>2</sub>, HCO<sub>3</sub>, pH e lactato);
- Parâmetros ventilatórios relacionados a VNI e CNAF (IPAP, EPAP, FiO<sub>2</sub>, fluxo de ar);
- Parâmetros relacionados ao paciente (Vt, FR e duração do tratamento em dias);
- Desfechos clínicos (taxa de necessidade de terapia de substituição renal, taxa de falha da VNI e/ou CNAF, tempo de internação hospitalar e na UTI, mortalidade intra-hospitalar);
- Serão registrados eventos adversos como: trombose venosa profunda, tromboembolismo pulmonar, acidente vascular encefálico, infarto agudo do miocárdio;

#### 3.7. Análise estatística:

Não houve cálculo de tamanho amostral devido à natureza exploratória, descritiva e retrospectiva deste estudo. Desta forma, todos os casos de março de 2020 à julho de 2021 serão considerados desde que tenham os critérios de inclusão e não tenham os critérios de exclusão. Para as estatísticas sumárias descritivas, as variáveis serão relatadas como média (desvio padrão), mediana (interquartil 25 – 75%) ou frequências absolutas e relativas, conforme apropriado.

O teste de U de Mann-Whitney será aplicado para avaliar diferenças no tempo de permanência da UTI. A estimativa de qualquer associação entre variáveis sobre os tipos de interface de suporte não invasivo (capacete, facial total, oronasal e CNAF), assim como os parâmetros ventilatórios utilizados será avaliada com análise univariada preliminar (teste qui-quadrado com correção de Yates ou teste exato de Fisher), seguida de modelo de regressão logística multivariada ajustado para todas as variáveis clínicas na admissão hospitalar. O tempo de sobrevivência, assim como tempo de internação hospitalar até o

evento serão analisados com estimativas de Kaplan-Meier; o teste de log-rank será utilizado para comparação entre grupos.

Os valores de p < 0,05 serão considerados estatisticamente significativos. Todas as análises serão realizadas utilizando-se SPSS® versão 25.0 (IBM Corp., Armonk, NY, USA).

## 4. ASPECTOS ÉTICOS E DE BOAS PRÁTICAS CLÍNICAS

Todo o estudo em seu planejamento, condução e publicação, será conduzido em conformidade com as boas práticas clínicas e as resoluções internacionais e nacionais relacionadas.

## 4.1. Aprovação do estudo:

O estudo foi aprovado pelo Comitê Cosubstanciado de Ética e Pesquisa do Instituto D'or de Pesquisa e Ensino, no dia 03 de Dezembro de 2021, sob número CAAE: 52534221.5.0000.5249.

## 5. DECLARAÇÃO DE CONFIDENCIALIDADE

Asseguramos que o sujeito de pesquisa incluído no estudo "FATORES PREDITIVOS PARA FALHA DA VENTILAÇÃO NÃO INVASIVA E DA OXIGENOTERAPIA SOB ALTO FLUXO EM PACIENTES COM COVID-19: ESTUDO OBSERVACIONAL RETROSPECTIVO" terá a sua confidencialidade resguardada pela equipe envolvida na condução do projeto de pesquisa e que, em nenhum momento, a identidade do paciente será revelada, conforme disposto na Res. CNS 466/12, item III. 2.i, e demais normas legislativas vigentes.

#### 6. ORÇAMENTO:

Os custos referentes à coleta de dados, produção do manuscrito e quaisquer outros decorrentes do projeto serão totalmente absorvidos pelos pesquisadores envolvidos.

## 7. CRONOGRAMA:

Protocolo: "FATORES PREDITIVOS PARA FALHA DA VENTILAÇÃO NÃO INVASIVA E DA OXIGENOTERAPIA SOB ALTO FLUXO EM PACIENTES COM COVID-19: ESTUDO OBSERVACIONAL RETROSPECTIVO"

| Atividades desenvolvidas | Início | Término | Local de realização |
|---|---|---|---|
| | | | da etapa |
| Aquisição de autorização para | 01/12/2021 | 20/12/2021 | Hospital Barra D'OR |
| acesso aos prontuários e | | | |
| treinamento para coleta de dados | | | |
| Levantamento de dados dos | 21/12/2021 | 21/05/2022 | Hospital Barra D'OR |
| prontuários eletrônicos | | | |
| Análise de dados preliminares e | 01/02/2022 | 09/03/2022 | Instituto de Biofísica |
| processo seletivo para o | | | Carlos Chagas Filho - |
| Mestrado | | | UFRJ |
| Ingresso ao Mestrado PPG | Março/2022 | Março/2024 | Instituto de Biofísica |
| (clínica médica) -UFRJ e | | | Carlos Chagas Filho - |
| realização de disciplinas | | | UFRJ |
| Organização dos dados obtidos | 22/05/2022 | 22/07/2022 | Instituto de Biofísica |
| dos prontuários eletrônicos | | | Carlos Chagas Filho - |
| | | | UFRJ |
| Análises estatísticas, inferências | 23/07/2022 | 23/09/2022 | Instituto de Biofísica |
| causais | | | Carlos Chagas Filho - |
| | | | UFRJ |
| Redação do manuscrito e | 24/09/2022 | 24/11/2022 | Instituto de Biofísica |
| submissão para revista científica | | | Carlos Chagas Filho - |
| | | | UFRJ |

#### 8. RESULTADOS PRELIMINARES

#### 8.1. Análise inicial

Conforme a coleta de dados se iniciou, foram reunidas e categorizadas as primeiras informações obtidas, primeiramente identificando os pacientes elegíveis para o estudo e categorizando-os nos grupos VNI, CNAF e VNI + CNAF (fase 1 da coleta de dados).

Na fase seguinte, a coleta de dados segue-se coletando os dados restantes prospostos na metodologia do estudo, reunindo, a princípio, apenas os dados de caracterização da população estudada no período proposto do estudo (fase 2 da coleta de dados).

As condições comorbidades, demográficas iniciais, e tempo de início dos sintomas dos grupos CNAF, VNI e VNI + CNAF foram reunidas e quantificadas na Tabela 1 e os resultados iniciais estão esquematizados no fluxograma a seguir.

**Tabela 1.** Condição demográfica inicial, comorbidades e tempo de sintomas conforme tratamentos utilizados

| | | | Trat | amentos | | | |
|---|---|---|---|---|---|---|---|
| | | CNAF | | VNI | VNI | + CNAF | |
| | N | col % | N | col % | N | col % | p-valor* |
| Não | 27 | 100,00% | 100 | 99,01% | 122 | 99,19% | 0,876 |
| Sim | 0 | 0,00% | 1 | 0,99% | 1 | 0,81% | |
| Não | 26 | 96,30% | 93 | 92,08% | 120 | 97,56% | 0,154 |
| Sim | 1 | 3,70% | 8 | 7,92% | 3 | 2,44% | |
| Não | 26 | 96,30% | 97 | 96,04% | 116 | 94,31% | 0,802 |
| Sim | 1 | 3,70% | 4 | 3,96% | 7 | 5,69% | |
| Não | 27 | 100,00% | 99 | 98,02% | 121 | 98,37% | 0,766 |
| Sim | 0 | 0,00% | 2 | 1,98% | 2 | 1,63% | |
| Não | 26 | 96,30% | 99 | 98,02% | 122 | 99,19% | 0,512 |
| Sim | 1 | 3,70% | 2 | 1,98% | 1 | 0,81% | |
| Não | 24 | 88,89% | 93 | 92,08% | 122 | 99,19% | 0,012 |
| Sim | 3 | 11,11% | 8 | 7,92% | 1 | 0,81% | |
| Não | 13 | 48,15% | 42 | 41,58% | 58 | 47,15% | 0,665 |
| Sim | 14 | 51,85% | 59 | 58,42% | 65 | 52,85% | |
| Não | 17 | 62,96% | 70 | 69,31% | 96 | 78,05% | 0,160 |
| Sim | 10 | 37,04% | 31 | 30,69% | 27 | 21,95% | |
| Não | 26 | 96,30% | 89 | 88,12% | 118 | 95,93% | 0,060 |
| Sim | 1 | 3,70% | 12 | 11,88% | 5 | 4,07% | |
| Não | 27 | 100,00% | 100 | 99,01% | 122 | 99,19% | 0,876 |
| | Sim Não Sim | N Não 27 Sim 0 Não 26 Sim 1 Não 26 Sim 1 Não 27 Sim 0 Não 26 Sim 1 Não 24 Sim 3 Não 13 Sim 14 Não 17 Sim 10 Não 26 Sim 1 | Não 27 100,00% Sim 0 0,00% Não 26 96,30% Sim 1 3,70% Não 26 96,30% Sim 1 3,70% Não 27 100,00% Sim 0 0,00% Não 26 96,30% Sim 1 3,70% Não 24 88,89% Sim 3 11,11% Não 13 48,15% Sim 14 51,85% Não 17 62,96% Sim 10 37,04% Não 26 96,30% Sim 1 3,70% | CNAF N col % N Não 27 100,00% 100 Sim 0 0,00% 1 Não 26 96,30% 93 Sim 1 3,70% 8 Não 26 96,30% 97 Sim 1 3,70% 4 Não 27 100,00% 99 Sim 0 0,00% 2 Não 26 96,30% 99 Sim 1 3,70% 2 Não 24 88,89% 93 Sim 3 11,11% 8 Não 13 48,15% 42 Sim 14 51,85% 59 Não 17 62,96% 70 Sim 10 37,04% 31 Não 26 96,30% 89 Sim 1 3,70% 12 | Não 27 100,00% 100 99,01% Sim 0 0,00% 1 0,99% Não 26 96,30% 93 92,08% Sim 1 3,70% 8 7,92% Não 26 96,30% 97 96,04% Sim 1 3,70% 4 3,96% Não 27 100,00% 99 98,02% Sim 0 0,00% 2 1,98% Não 26 96,30% 99 98,02% Sim 1 3,70% 2 1,98% Não 24 88,89% 93 92,08% Sim 3 11,11% 8 7,92% Não 13 48,15% 42 41,58% Sim 14 51,85% 59 58,42% Não 17 62,96% 70 69,31% Sim 10 37,04% 31 30,69% | CNAF VNI VNI N col % N col % N Não 27 100,00% 100 99,01% 122 Sim 0 0,00% 1 0,99% 1 Não 26 96,30% 93 92,08% 120 Sim 1 3,70% 8 7,92% 3 Não 26 96,30% 97 96,04% 116 Sim 1 3,70% 4 3,96% 7 Não 27 100,00% 99 98,02% 121 Sim 0 0,00% 2 1,98% 2 Não 26 96,30% 99 98,02% 122 Sim 1 3,70% 2 1,98% 1 Não 24 88,89% 93 92,08% 122 Sim 3 11,11% 8 7,92% 1 Não 13 48,15% < | CNAF VNI VNI + CNAF Não 27 100,00% 100 99,01% 122 99,19% Sim 0 0,00% 1 0,99% 1 0,81% Não 26 96,30% 93 92,08% 120 97,56% Sim 1 3,70% 8 7,92% 3 2,44% Não 26 96,30% 97 96,04% 116 94,31% Sim 1 3,70% 4 3,96% 7 5,69% Não 27 100,00% 99 98,02% 121 98,37% Sim 0 0,00% 2 1,98% 2 1,63% Não 26 96,30% 99 98,02% 122 99,19% Sim 1 3,70% 2 1,98% 1 0,81% Não 26 96,30% 99 98,02% 122 99,19% Sim 1 3,70% <td< td=""></td<> |

| Paciente Sim imunossuprimidos | | 0 | 0,00% | 1 | 0,99% | 1 | 0,81% | |
|---|---|---|---|---|---|---|---|---|
| Obesidade | Não | 16 | 59,26% | 67 | 66,34% | 72 | 58,54% | 0,470 |
| | Sim | 11 | 40,74% | 34 | 33,66% | 51 | 41,46% | |
| Demência | Não | 27 | 100,00% | 94 | 93,07% | 122 | 99,19% | 0,021 |
| | Sim | 0 | 0,00% | 7 | 6,93% | 1 | 0,81% | |
| Outras Comorbidades | Não | 15 | 55,56% | 39 | 38,61% | 61 | 49,59% | 0,146 |
| | Sim | 12 | 44,44% | 62 | 61,39% | 62 | 50,41% | |
| Gênero | F | 8 | 29,63% | 32 | 31,68% | 30 | 24,39% | 0,470 |
| | M | 19 | 70,37% | 69 | 68,32% | 93 | 75,61% | |
| Tempo de sintomas | 0 a 10 dias | 14 | 77,78% | 51 | 98,08% | 65 | 94,20% | 0,037 |
| | 11 a 20 dias | 3 | 16,67% | 1 | 1,92% | 2 | 2,90% | |
| | 21 a 30 dias | 1 | 5,55% | 0 | 0,00% | 2 | 2,90% | |
| | Mais de 30 dias | 0 | 0,00% | 0 | 0,00% | 0 | 0,00% | |
| Idade | 16 a 39 anos | 1 | 3,70% | 12 | 12,37% | 19 | 15,57% | 0,002 |
| | 40 a 59 anos | 9 | 33,33% | 35 | 36,08% | 56 | 45,90% | |
| | 60 a 79 anos | 14 | 51,85% | 30 | 30,93% | 44 | 36,07% | |
| | 80 a 99 anos | 3 | 11,11% | 19 | 19,59% | 3 | 2,46% | |
| | 100 anos ou mais | 0 | 0,00% | 1 | 1,03% | 0 | 0,00% | |
| Índice de Massa Corpórea (IMC) | IMC maior ou igual a 30 | 11 | 61,11% | 23 | 50,00% | 38 | 49,35% | 0,658 |
| . , | IMC menor que 30 | 7 | 38,89% | 23 | 50,00% | 39 | 50,65% | |
| *Teste de qui quadrado | | | | | | | | |

O tempo de início dos sintomas está demonstrado na Tabela 2. Não há diferença entre os tratamentos VNI, CNAF e VNI + CNAF (Tabela 2). A ausência de cardiopatia e demência, assim como o início dos sintomas menor ou igual à 10 dias e a idade destacam-se, inicialmente, com relação à adoção da terapia instalada (Figuras 3, 4). A instalação da VNI e/ou CNAF na fase aguda da doença (primeiros 10 dias de sintomas) predomina em todos os grupos estudados até o momento (Figura 5), enquanto que a faixa etária entre 40 e 79 anos constitui o principal grupo submetido à VNI e/ou CNAF.

Tabela 2. Tempo de sintomas e IMC conforme tratamentos utilizados

| | | Tratamentos | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Só CNAF | (n=27) | | Só VNI (n=101) | | | | VNI + CNAF (n=123) | | | |
| Variável | M | MD | DP | IIQ | M | MD | DP | IIQ | M | MD | DP | IIQ |
| Tempo de sintomas (dias) | 7,22 | 6 | 6,11 | 5,5 | 4,23 | 4 | 3,1 | 4 | 4,99 | 4 | 4,72 | 2 |

M: média; MD: mediana; DP: desvio padrão; IIQ: O intervalo interquartil.

Figura 3. Cardiopatia ou não conforme tratamentos



Figura 4. Demência ou não conforme tratamentos



Figura 5. Tempo de sintomas conforme tratamentos



Figura 6. Faixa etária conforme tratamentos

#### ANEXO 1: FLUXOGRAMA DOS DADOS PRELIMINARES



<sup>\*</sup> A partir dos 1090 prontuários avaliados até o momento.

<sup>\*\*</sup> Os prontuários avaliados até o momento ainda não passaram pelos critérios de exclusão

### 9. REFERÊNCIAS BIBLIOGRÁFICAS

ACKERMANN, M. et al. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. **New England Journal of Medicine**, v. 383, n. 2, p. 120–128, 9 jul. 2020.

ALBARELLO, F. et al. 2019-novel Coronavirus severe adult respiratory distress syndrome in two cases in Italy: An uncommon radiological presentation. **International Journal of Infectious Diseases**, v. 93, p. 192–197, abr. 2020.

ALRADDADI, B. M. et al. Noninvasive ventilation in critically ill patients with the Middle East respiratory syndrome. **Influenza and Other Respiratory Viruses**, v. 13, n. 4, p. 382–390, jul. 2019.

BATISTA, A. et al. Análise socioeconômica da taxa de letalidade da COVID-19 no Brasil. p. 12, [s.d.].

BATTAGLINI, D. et al. Noninvasive respiratory support and patient self-inflicted lung injury in COVID-19: a narrative review. **British Journal of Anaesthesia**, v. 127, n. 3, p. 353–364, set. 2021.

BERLIN, D. A.; GULICK, R. M.; MARTINEZ, F. J. Severe Covid-19. **New England Journal of Medicine**, v. 383, n. 25, p. 2451–2460, 17 dez. 2020a.

BERLIN, D. A.; GULICK, R. M.; MARTINEZ, F. J. Severe Covid-19. **New England Journal of Medicine**, v. 383, n. 25, p. 2451–2460, 17 dez. 2020b.

BERTAINA, M. et al. Non-invasive ventilation for SARS-CoV-2 acute respiratory failure: a subanalysis from the HOPE COVID-19 registry. **Emergency Medicine Journal**, v. 38, n. 5, p. 359–365, maio 2021.

BOCCHILE, R. L. R. et al. The effects of high-flow nasal cannula on intubation and reintubation in critically ill patients: a systematic review, meta-analysis and trial sequential analysis. **Revista Brasileira de Terapia Intensiva**, v. 30, n. 4, 2018.

BOGOCH, I. I. et al. Pneumonia of unknown aetiology in Wuhan, China: potential for international spread via commercial air travel. **Journal of Travel Medicine**, v. 27, n. 2, p. taaa008, 13 mar. 2020.

CARVALHO, A. R. S. et al. Estimating COVID-19 Pneumonia Extent and Severity From Chest Computed Tomography. **Frontiers in Physiology**, v. 12, p. 617657, 15 fev. 2021.

R Core Team: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/. 2021.

CRUCES, P. et al. A physiological approach to understand the role of respiratory effort in the progression of lung injury in SARS-CoV-2 infection. **Critical Care**, v. 24, n. 1, p. 494, dez. 2020.

Diretrizes\_Brasileiras\_de\_Ventilacao\_Mecanica\_2013\_AMIB\_SBPT\_Arquivo\_Eletronico Oficial.pdf., [s.d.].

FERREYRO, B. L. et al. Association of Noninvasive Oxygenation Strategies With All-Cause Mortality in Adults With Acute Hypoxemic Respiratory Failure: A Systematic Review and Meta-analysis. **JAMA**, v. 324, n. 1, p. 57, 7 jul. 2020.

FRANCO, C. et al. Feasibility and clinical impact of out-of-ICU noninvasive respiratory support in patients with COVID-19-related pneumonia. **European Respiratory Journal**, v. 56, n. 5, p. 2002130, nov. 2020.

GATTINONI, L. et al. COVID-19 pneumonia: different respiratory treatments for different phenotypes? **Intensive Care Medicine**, v. 46, n. 6, p. 1099–1102, jun. 2020.

GATTINONI, L.; CARLESSO, E.; CAIRONI, P. Stress and strain within the lung: **Current Opinion in Critical Care**, v. 18, n. 1, p. 42–47, fev. 2012.

GRIECO, D. L. et al. Patient self-inflicted lung injury: implications for acute hypoxemic respiratory failure and ARDS patients on non-invasive support. **Minerva Anestesiologica**, v. 85, n. 9, set. 2019.

HANI, C. et al. COVID-19 pneumonia: A review of typical CT findings and differential diagnosis. **Diagnostic and Interventional Imaging**, v. 101, n. 5, p. 263–268, maio 2020.

HOFFMANN, M. et al. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. **Cell**, v. 181, n. 2, p. 271-280.e8, abr. 2020.

JAMILLOUX, Y. et al. Should we stimulate or suppress immune responses in COVID-19? Cytokine and anti-cytokine interventions. **Autoimmunity Reviews**, v. 19, n. 7, p. 102567, jul. 2020.

KURTZ, P. et al. Envolving changes in mortality of 13,301 critically ill adult patients with COVID-19 over 8 months. Intensive Care Medicine, v 47, p. 538–548, 2021.

LIN, L. et al. Hypothesis for potential pathogenesis of SARS-CoV-2 infection—a review of immune changes in patients with viral pneumonia. **Emerging Microbes & Infections**, v. 9, n. 1, p. 727–732, 1 jan. 2020.

LOPES-PACHECO, M. et al. Pathogenesis of Multiple Organ Injury in COVID-19 and Potential Therapeutic Strategies. **Frontiers in Physiology**, v. 12, p. 593223, 28 jan. 2021.

MALIK, Y. S. et al. Coronavirus Disease Pandemic (COVID-19): Challenges and a Global Perspective. **Pathogens**, v. 9, n. 7, p. 519, 28 jun. 2020.

MANCIA, G. et al. Renin-Angiotensin-Aldosterone System Blockers and the Risk of Covid-19. **New England Journal of Medicine**, v. 382, n. 25, p. 2431–2440, 18 jun. 2020.

MENG, L. et al. Intubation and Ventilation amid the COVID-19 Outbreak. **Anesthesiology**, v. 132, n. 6, p. 1317–1332, 1 jun. 2020.

MENGA, L. S. et al. High Failure Rate of Noninvasive Oxygenation Strategies in Critically Ill Subjects With Acute Hypoxemic Respiratory Failure Due to COVID-19. **Respiratory Care**, v. 66, n. 5, p. 705–714, maio 2021.

NISHIMURA, M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. **Respiratory Care**, v. 61, n. 4, p. 529–541, 1 abr. 2016.

Postmortem Examination of Patients With COVID-19. p. 3, 2020.

RADOVANOVIC, D. et al. Mortality and clinical outcomes in patients with COVID-19 pneumonia treated with non-invasive respiratory support: A rapid review. **Journal of Critical Care**, v. 65, p. 1–8, out. 2021.

RANZANI, O. T. Characterisation of the first 250 000 hospital admissions for COVID-19 in Brazil: a retrospective analysis of nationwide data. p. 12, [s.d.].

RELLO, J. et al. Clinical phenotypes of SARS-CoV-2: implications for clinicians and researchers. **European Respiratory Journal**, v. 55, n. 5, p. 2001028, maio 2020.

RISC-19-ICU INVESTIGATORS et al. Implications of early respiratory support strategies on disease progression in critical COVID-19: a matched subanalysis of the prospective RISC-19-ICU cohort. **Critical Care**, v. 25, n. 1, p. 175, dez. 2021.

ROBBA, C. et al. Distinct phenotypes require distinct respiratory management strategies in severe COVID-19. **Respiratory Physiology & Neurobiology**, v. 279, p. 103455, ago. 2020.

ROBBA, C. et al. Coagulative Disorders in Critically Ill COVID-19 Patients with Acute Distress Respiratory Syndrome: A Critical Review. **Journal of Clinical Medicine**, v. 10, n. 1, p. 140, 3 jan. 2021.

ROCHWERG, B. et al. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. **European Respiratory Journal**, v. 50, n. 2, p. 1602426, ago. 2017.

RODRIGUEZ-MORALES, A. J. et al. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. **Travel Medicine and Infectious Disease**, v. 34, p. 101623, mar. 2020.

SIDDIQI, H. K.; MEHRA, M. R. COVID-19 illness in native and immunosuppressed states: A clinical—therapeutic staging proposal. **The Journal of Heart and Lung Transplantation**, v. 39, n. 5, p. 405–407, maio 2020.

SLUTSKY, A. S.; RANIERI, V. M. Ventilator-Induced Lung Injury. **New England Journal of Medicine**, v. 369, n. 22, p. 2126–2136, 28 nov. 2013.

TAHAMTAN, A.; ARDEBILI, A. Real-time RT-PCR in COVID-19 detection: issues affecting the results. **Expert Review of Molecular Diagnostics**, v. 20, n. 5, p. 453–454, 3 maio 2020.

TAY, M. Z. et al. The trinity of COVID-19: immunity, inflammation and intervention. **Nature Reviews Immunology**, v. 20, n. 6, p. 363–374, jun. 2020.

UZUNIAN, A. Coronavirus SARS-CoV-2 and Covid-19. **Jornal Brasileiro de Patologia e Medicina Laboratorial**, 2020.

VABRET, N. et al. Immunology of COVID-19: Current State of the Science. **Immunity**, v. 52, n. 6, p. 910–941, jun. 2020.

VOM ELM, E. et. al. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: Guidelines for Reporting Observational Studies. PLoS Med 4(10): e296, 2007

WEERAKKODY, S. et al. Non-invasive respiratory support in the management of acute COVID-19 pneumonia: considerations for clinical practice and priorities for research. **The Lancet Respiratory Medicine**, p. S2213260021004148, nov. 2021.

XU, X.-P. et al. Noninvasive Ventilation in Acute Hypoxemic Nonhypercapnic Respiratory Failure: A Systematic Review and Meta-Analysis. **Critical Care Medicine**, v. 45, n. 7, p. e727–e733, jul. 2017.

YOSHIDA, T. et al. Spontaneous Effort Causes Occult Pendelluft during Mechanical Ventilation. **American Journal of Respiratory and Critical Care Medicine**, v. 188, n. 12, p. 1420–1427, 15 dez. 2013.

ZARRILLI, G. et al. The Immunopathological and Histological Landscape of COVID-19-Mediated Lung Injury. **International Journal of Molecular Sciences**, v. 22, n. 2, p. 974, 19 jan. 2021.

https://www.paho.org/pt/brasil - acesso em 14 de dezembro de 2021.

https://www.who.int/ - acesso em 14 de dezembro de 2021.

https://covid.saude.gov.br/ - acesso em 14 de dezembro de 2021.

https://ourworldindata.org/covid-vaccinations?country=BRA - acesso em 14 de dezembro de 2021.

https://www.ufrgs.br/coronaviruslitoral/uma-breve-linha-do-tempo/ - acesso em 14 de dezembro de 2021.